CLINICAL TRIAL: NCT06883422
Title: Impact of Pre-surgical Oral Immunonutrition on Plasma Levels of Branched-chain Amino Acids in Elective Colorectal Surgery Patients: a Randomized, Double-blind, Controlled, Clinical Trial
Brief Title: Pre-Surgical Immunonutrition's Effect on Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Aurora Elizabeth Serralde Zúñiga, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4475
Record Dates: First submitted 2025-03-07; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Surgery
Keywords: Colorectal Surgery; Immunonutrition; Enhanced Recovery After Surgery; Preoperative Care; Amino Acids Branched-Chain

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled clinical trial
  Sample Size:
  For the sample size calculation, it was considered that patients in the immunonutrition intervention group will have a 21% increase in plasma branched-chain amino acid concentration, as reported in the study by Cangiano C et al. Therefore, considering a type 1 error (α) of 0.05 with one tail, and a type 2 error (β) of 0.20, and using the formula N = 2s² (Zα + Zβ)² / Δ², a sample size of 63 subjects per group is obtained.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Preoperative oral supplementation (immunonutrition)
  Interventions: Dietary Supplement: Preoperative oral immunonutrition formula
- Control Arm (Active Comparator): Preoperative oral supplementation (polymeric)
  Interventions: Dietary Supplement: Preoperative oral Isocaloric and isoproteic polymeric formula

INTERVENTIONS:
Dietary Supplement: Preoperative oral immunonutrition formula — Intervention arm will daily receive, for 7 days, a preoperative oral formula with immunonutrients: 500 kcal of energy, 41 g of protein, 60 g of carbohydrates, 11 g of lipids, 5.7 g of glutamine, 7 g of arginine, 3.6 g of leucine, 2.7 g of isoleucine, 3.7 g of valine, and 0.35 g of omega 3
  Arms: Intervention Arm
Dietary Supplement: Preoperative oral Isocaloric and isoproteic polymeric formula — Control arm will daily receive, for 7 days, an isocaloric and isoproteic preoperative oral formula: 500 kcal of energy, 41 g of protein, 60 g of carbohydrates, and 11 g of lipids
  Arms: Control Arm

SUMMARY:
Colorectal surgery patients face excessive catabolism, increasing inflammation and immune compromise. The administration of nutritional supplements known as immunonutrition before gastrointestinal surgery has been shown to improve clinical outcomes; however, the mechanisms underlying these benefits remain inconclusive.

The objective of the study is to evaluate the effect of preoperative nutritional supplementation with an immunonutrient-enriched formula compared to an isocaloric and isoproteic formula on plasma BCAA concentration in patients undergoing elective colorectal surgery. A double-blind, randomized controlled clinical trial will be conducted. Patients will be required to drink the supplement daily for the 7 days preceding the surgical intervention. Patients in both groups will be instructed to maintain their usual food intake. During the study, there will be two patient assessments and a review of medical records to document the outcomes.

DETAILED DESCRIPTION:
Patients undergoing colorectal surgery, experience excessive and persistent catabolism, leading to skeletal muscle depletion, and increased inflammatory and immunological involvement, this results in greater malnutrition, mortality, and postoperative morbidity. Depletion of amino acids leads to an increased inflammatory response and diminished immunity. Guidelines of leading international societies in the field of clinical nutrition recommend the perioperative administration of oral formulas with immunonutrients in these patients. The administration of nutritional supplements known as immunonutrition (fortified with arginine, glutamine, branched-chain amino acids (BCAAs) and omega-3 polyunsaturated fatty acids) before gastrointestinal surgery has been shown to improve clinical outcomes, such as a reduction in post-surgical infectious, reduced risk of anastomotic leakage and fewer days of hospital stay; however, the mechanisms related to these benefits are not conclusive.

The aim of the study is to evaluate the effect of preoperative nutritional supplementation for 7 days with a formula enriched with immunonutrients compared to an isocaloric and isoproteic formula, on the plasma concentration of BCAAs in patients undergoing elective colorectal surgery. A randomized, double-blind, controlled trial will be conducted with 63 patients per group. The concentration of BCAAs will be measured prior to the 7 days of nutritional supplementation and will be repeated on the day of the surgical intervention before the procedure. The supplements for both groups will provide 500 calories, 41 g of protein, 60 g of carbohydrates, and 11 g of lipids; the supplement for the intervention group is additionally fortified with immunonutrients. Patients will be instructed to consume the supplement daily for the 7 days prior to the surgical intervention. Patients in both groups will be advised to maintain their usual food intake.

The investigators hypothesized that if an oral formula with immunonutrients is administered compared to an isocaloric and isoproteic formula without them for 7 days in the preoperative period in patients undergoing elective colorectal surgery, there will be an increase in the plasma concentration of BCAAs in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Over 18 years of age
* Scheduled for elective colorectal surgery (Resection and intestinal reconnection)
* Obtaining patient consent

Exclusion Criteria:

* Consumption of nutritional supplements during the 2 weeks prior to patient enrollment
* Consumption of additional nutritional supplements during the 7 days corresponding to the study intervention period
* Patients diagnosed with chronic kidney disease
* Patients diagnosed with hepatic cirrhosis
* Documented allergy to any of the ingredients in the formulas under evaluation (milk and/or soy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of branched-chain amino acids | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement). The second measurement will be performed on the day of the surgical intervention, before the start of the procedure
  Plasma concentrations of branched-chain amino acids, expressed in micromoles per liter (µmol/L), will be quantified at two distinct time points during the study

SECONDARY OUTCOMES:
Concentration of albumin | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement). The second measurement will be performed on the day of the surgical intervention, before the start of the procedure
  Serum concentrations of albumin, expressed in grams per deciliter (g/dL), will be quantified at two distinct time points during the study
Concentration of high-sensitivity C-reactive protein | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement). The second measurement will be performed on the day of the surgical intervention, before the start of the procedure
  Serum concentrations of high-sensitivity C-reactive protein, expressed in milligrams per deciliter (mg/dL), will be quantified at two distinct time points during the study
Mortality | Mortality will be assessed within 30 days post-surgery
  The incidence of death within the study population will be recorded and reported throughout the study period following surgery
Length of stay | Length of stay will be assessed within 30 days post-surgery
  The number of days from the patient's hospital admission to discharge will be recorded and reported during the study period
Hospital readmission | Hospital readmission will be assessed within 30 days post-surgery
  The necessity for rehospitalization after discharge following surgery will be recorded and reported during the study period
Anastomotic dehiscence | Anastomotic dehiscence will be assessed within 30 days post-surgery
  Occurrence of anastomotic dehiscence within the study population following surgery
Surgical site infection | Surgical site infection will be assessed within 30 days post-surgery
  Occurrence of surgical site infection within the study population following surgery
Fistula | Fistula will be assessed within 30 days post-surgery
  Occurrence of fistula within the study population following surgery
Paralytic ileus | Paralytic ileus will be assessed within 30 days post-surgery
  Occurrence of paralytic ileus within the study population following surgery
Postoperative intestinal obstruction | Postoperative intestinal obstruction will be assessed within 30 days post-surgery
  Occurrence of postoperative intestinal obstruction within the study population following surgery

OTHER OUTCOMES:
Weight | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Weight will be measured using a calibrated scale and quantified at two distinct time points during the study and will be reported in kg
Height | The measurement will be conducted 7 days prior to the surgical intervention
  Height will be assessed using a standardized automatic stadiometer and quantified once during the study and will be reported in cm
Body mass index | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Body mass index (BMI) will be calculated from the measured weight and height, quantified at two distinct time points during the study and will be reported in kg/m2
Muscle mass | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Muscle mass will be evaluated using a standardized tetrapolar bioelectrical impedance analysis and quantified at two distinct time points during the study and will be reported in % of the body weight
Fat mass | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Fat mass will be evaluated using a standardized tetrapolar bioelectrical impedance analysis and quantified at two distinct time points during the study and will be reported in % of the body weight
Phase angle | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Phase angle will be evaluated using a standardized tetrapolar bioelectrical impedance analysis and quantified at two distinct time points during the study and will be reported in degrees (°)
Muscle strength | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Muscle strength will be measured in the dominant hand using a hand dynamometer following a standardized protocol and quantified at two distinct time points during the study and will be reported in kg
Calf circumference | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Calf circumference will be measured using a standardized, non-stretchable metallic tape with standard anthropometric techniques and quantified at two distinct time points during the study and will be reported in cm
Mid-arm circumference | The first measurement will be conducted 7 days prior to the surgical intervention (baseline measurement), and the second measurement will be performed on the day of the surgical intervention before the procedure begins
  Mid-arm circumference will be measured using a standardized, non-stretchable metallic tape with standard anthropometric techniques and quantified at two distinct time points during the study and will be reported in cm
Abdominal distension | The assessment will be conducted on the day of the surgical intervention before the procedure begins.
  Abdominal distension will be recorded through patient self-report and will be reported as presence or absence
Abdominal pain | The assessment will be conducted on the day of the surgical intervention before the procedure begins
  Abdominal pain will be recorded through patient self-report and will be reported as presence or absence
Diarrhea | The assessment will be conducted on the day of the surgical intervention before the procedure begins
  The occurrence of diarrhea will be recorded through patient self-report and will be reported as presence or absence
Nausea | The assessment will be conducted on the day of the surgical intervention before the procedure begins
  The occurrence of nausea will be recorded through patient self-report and will be reported as presence or absence
Vomiting | The assessment will be conducted on the day of the surgical intervention before the procedure begins
  The occurrence of vomiting will be recorded through patient self-report and will be reported as presence or absence

CONTACTS AND LOCATIONS:
Overall Officials: Aurora E Serralde Zúñiga, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Aurora E Serralde Zúñiga, MD, PhD, Mexico City, Tlalpan, Mexico

REFERENCES:
- [Background] Li P, Yin YL, Li D, Kim SW, Wu G. Amino acids and immune function. Br J Nutr. 2007 Aug;98(2):237-52. doi: 10.1017/S000711450769936X. Epub 2007 Apr 3. PMID 17403271
- [Background] Choudry HA, Pan M, Karinch AM, Souba WW. Branched-chain amino acid-enriched nutritional support in surgical and cancer patients. J Nutr. 2006 Jan;136(1 Suppl):314S-8S. doi: 10.1093/jn/136.1.314S. PMID 16365105
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Finco C, Magnanini P, Sarzo G, Vecchiato M, Luongo B, Savastano S, Bortoliero M, Barison P, Merigliano S. Prospective randomized study on perioperative enteral immunonutrition in laparoscopic colorectal surgery. Surg Endosc. 2007 Jul;21(7):1175-9. doi: 10.1007/s00464-007-9238-4. Epub 2007 Mar 14. PMID 17356942
- [Background] Slim K, Badon F, Vacheron CH, Dziri C, Marquillier T. Efficacy of perioperative immunonutrition in visceral surgery: an umbrella review protocol. BMJ Open. 2021 Sep 13;11(9):e053851. doi: 10.1136/bmjopen-2021-053851. PMID 34518277
- [Background] Adiamah A, Skorepa P, Weimann A, Lobo DN. The Impact of Preoperative Immune Modulating Nutrition on Outcomes in Patients Undergoing Surgery for Gastrointestinal Cancer: A Systematic Review and Meta-analysis. Ann Surg. 2019 Aug;270(2):247-256. doi: 10.1097/SLA.0000000000003256. PMID 30817349
- [Background] Yu K, Zheng X, Wang G, Liu M, Li Y, Yu P, Yang M, Guo N, Ma X, Bu Y, Peng Y, Han C, Yu K, Wang C. Immunonutrition vs Standard Nutrition for Cancer Patients: A Systematic Review and Meta-Analysis (Part 1). JPEN J Parenter Enteral Nutr. 2020 Jul;44(5):742-767. doi: 10.1002/jpen.1736. Epub 2019 Nov 11. PMID 31709584
- [Background] Niu JW, Zhou L, Liu ZZ, Pei DP, Fan WQ, Ning W. A Systematic Review and Meta-Analysis of the Effects of Perioperative Immunonutrition in Gastrointestinal Cancer Patients. Nutr Cancer. 2021;73(2):252-261. doi: 10.1080/01635581.2020.1749291. Epub 2020 Apr 14. PMID 32285694
- [Background] Cangiano C, Laviano A, Meguid MM, Mulieri M, Conversano L, Preziosa I, Rossi-Fanelli F. Effects of administration of oral branched-chain amino acids on anorexia and caloric intake in cancer patients. J Natl Cancer Inst. 1996 Apr 17;88(8):550-2. doi: 10.1093/jnci/88.8.550. No abstract available. PMID 8606384